CLINICAL TRIAL: NCT07385469
Title: Effects of the Sequential Oral Sensory Feeding Approach and Occupational Performance Coaching in Children With Avoidant/Restrictive Food Intake Disorder (ARFID): A Randomized Controlled Trial
Brief Title: Sensory Feeding and Parent Coaching for Children With ARFID
Acronym: SOS OPC ARFID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ezginur Gündoğmuş, Research assisstant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SBF 25/092
Record Dates: First submitted 2025-09-05; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: ARFID
Keywords: ARFID; Eating Disorder; Occupational Therapy; Sensory Feeding; Occupational Performance Coaching
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: This randomized, single-blind, controlled study will be conducted with children aged 3-8 years who were diagnosed with ARFID by a Child and Adolescent Psychiatrist according to DSM-V criteria and referred to the occupational therapy department. Based on the power analysis using effect size (f = 0.35), α = 0.05, and power (1-β) = 0.80, a total of 39 children were required, with at least 13 participants in each group. With a 15% probability of missing data estimate, the total sample size was determined to be 45 children. The Consort checklist used for randomized controlled trials will be used in the study design. The single-blind method in the study is based on the principle that the experts conducting the evaluations are unaware of the group assignment; thus, the measurement results will be evaluated independently of any knowledge of the intervention. While the intervention providers have knowledge of the groups, the analysts will work blindly during the data analysis phase. Informed co
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The single-blind method in this study is based on the principle that the experts conducting the evaluations are unaware of the group assignment; thus, the measurement results will be evaluated independently of the intervention information. While the intervention implementers have knowledge of the groups, analysts during the data analysis phase will be blinded to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The group that applied only the SOS approach for 60 minutes, once a week for 12 weeks (Active Comparator): Children in the first group will receive the intervention once a week for 60 minutes over a period of 12 weeks. The SOS approach is used as a structured intervention that supports sensory-motor skills related to feeding and aims to help the child develop a positive relationship with food. By gradually increasing interaction with food, the SOS approach aims to reduce sensory sensitivities and improve feeding behaviors. The intervention is structured to increase the child's tolerance to food through the following sequence:
  Visual Tolerance
  The child only looks at the food without physical contact.
  The food remains on the table, maintaining distance from the child.
  Phrases such as "we can just look at this" or "we can recognize it with our eyes" are used.
  Bringing Food Closer / Smelling
  The food is brought into the child's personal space.
  To build tolerance to smell, the food is held close to the nose.
  This stage is particularly important for children with olfactory sensitivities
  Interventions: Behavioral: Sequential Oral Sensory (SOS) Feeding Approach
- The group that received 60 minutes of SOS + 30 minutes of OPC once a week for 12 weeks (Active Comparator): Children in the second group will receive the SOS approach combined with the Occupational Performance Coaching (OPC) program. After completing the 60-minute SOS session, 30-minute OPC sessions will also be delivered once a week for 12 weeks on an individual basis.
  OPC enables parents to set goals, develop strategies, and evaluate progress aimed at improving their child's daily life performance.
  Sessions are conducted in a semi-structured interview format with the therapist.
  Focus areas include: establishing feeding routines, parent-child interaction, home-based implementation strategies, and parental self-efficacy.
  OPC is a family-centered, occupation-based, coaching approach implemented by occupational therapists in collaboration with families to enhance children's participation in daily life. The aim is to guide parents in making environmental adjustments that support their children's functional goals and to empower them to generate their own solutions.
  Phases of OPC:
  Goal Set
  Interventions: Behavioral: SOS + Occupational Performance Coaching (OPC)
- Control Group (Waitlist) (No Intervention): Participants assigned to the control group will be placed on a waiting list and will not receive any intervention during the 12-week study period. They will complete baseline and post-test assessments at the same time points as the intervention groups, allowing for comparison of outcomes. After the study is completed, families in this group will be offered the effective intervention program outside of the research protocol to ensure ethical access to treatment.

INTERVENTIONS:
Behavioral: Sequential Oral Sensory (SOS) Feeding Approach — The SOS Feeding Approach is a structured, evidence-informed intervention that gradually exposes children with ARFID to food across multiple sensory dimensions, recognizing that these children often experience heightened sensitivities to textures, smells, and tastes that can trigger avoidance and distress. Unlike traditional behavioral methods that focus primarily on intake, SOS emphasizes building comfort, positive associations, and sensory tolerance before progressing to consumption. Delivered in 12 weekly 60-minute sessions by trained occupational therapists, the approach is individualized to each child's developmental stage, medical history, and swallowing safety, with foods selected accordingly. Sessions progress through a hierarchy-visual tolerance, olfactory exposure, tactile exploration, oral contact, intraoral exploration, and finally chewing and swallowing-ensuring gradual, non-coercive acceptance. By integrating sensory-motor learning with feeding, the intervention reduces m
  Arms: The group that applied only the SOS approach for 60 minutes, once a week for 12 weeks
Behavioral: SOS + Occupational Performance Coaching (OPC) — In the combined SOS and OPC intervention, children receive a 60-minute SOS session each week for 12 weeks, immediately followed by a 30-minute OPC session with their parents. SOS targets the child's sensory tolerance and positive engagement with food, while OPC uses a semi-structured coaching format where parents set meaningful feeding goals, analyze mealtime routines, and develop sustainable strategies with the therapist. Parents implement these strategies at home and review progress in subsequent sessions, ensuring continuous feedback and adjustment. This dual approach is distinguished by its family-centered nature, empowering parents as active agents of change, and by its integration of child-focused sensory therapy with parent coaching to reinforce improvements across home and clinical settings. By addressing both sensory challenges and parent-child dynamics, the intervention aims to reduce mealtime anxiety, expand food acceptance, strengthen parental self-efficacy, and achieve mor
  Arms: The group that received 60 minutes of SOS + 30 minutes of OPC once a week for 12 weeks

SUMMARY:
This study aims to investigate the effects of the SOS approach alone, or the SOS approach plus the OPC intervention, on children's feeding problems and feeding behaviors, as well as parents' feeding attitudes and mealtime behaviors in children diagnosed with ARFID. This randomized, single-blind, controlled trial will be conducted with children aged 3-8 years who were diagnosed with ARFID by a Child and Adolescent Psychiatrist according to DSM-V criteria and referred to an occupational therapy department. Power analysis determined the sample size to be 45 children (15 per group). Participants will be assigned to three groups using computer-assisted block randomization: Group 1: Sequential Oral Sensory (SOS) Feeding Approach alone; Group 2: SOS approach plus Occupational Performance Coaching (OPC); and Group 3: Control group (standard follow-up without intervention). The study design will utilize the Consort checklist used for randomized controlled trials. Informed consent will be obtained from participants. Pre- and post-intervention assessments will be conducted on the child's feeding behaviors, food variety, and mealtime negative behaviors, as well as parental feeding attitudes, mealtime behaviors, and stress. The study concludes that feeding interventions implemented using the SOS approach will be effective in reducing food acceptance, food variety, and mealtime negative behaviors in children with ARFID. These effects are expected to be more pronounced and sustained when Occupational Performance Coaching (OPC) is added to the SOS approach. Furthermore, positive changes in parents' feeding attitudes and strengthened parent-child interactions at mealtime are anticipated. These results will contribute to the literature on the effectiveness of using sensory-based approaches and family-based counseling in combination in interventions for ARFID. They are also expected to provide an evidence-based roadmap for occupational therapists to develop holistic intervention programs when working with children with ARFID in clinical practice.

DETAILED DESCRIPTION:
Avoidant/Restrictive Food Intake Disorder (ARFID), defined and included in the diagnostic categories with the publication of the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) by the American Psychiatric Association, is a serious disorder related to feeding behavior. According to DSM-5, ARFID is characterized by one or more of the following criteria: significant weight loss (or failure to achieve expected weight gain/growth in children), marked nutritional deficiencies, dependence on enteral feeding or oral nutritional supplements, and/or marked impairment in psychosocial functioning. This condition differs from culturally normative fasting or attempts to lose weight and is not associated with a fear of body shape or weight.

In children with ARFID, food selectivity, insufficient food intake, and intense negative emotions related to feeding are observed. This disorder not only leads to weight loss and growth retardation but also significantly affects children's daily life activities, family life, and social interactions.

ARFID has a prevalence rate of 3.2% in the general pediatric population. It has been reported that the proportion of males is higher in ARFID diagnoses and that, compared to other DSM-5 eating disorders, it is more frequently associated with comorbid psychiatric and/or medical conditions. However, ARFID is a heterogeneous condition that includes individuals ranging from young children to adults. Prevalence estimates for ARFID vary widely depending on the population and setting examined. A systematic review found that in non-clinical child and adolescent samples, estimated prevalence rates for ARFID ranged between 0.3% and 15.5%. The prevalence has been reported as 64% among infants and young children, and 15.5% among children aged 5-10 years.

To date, most research on ARFID treatment has focused on psychological interventions, which typically include psychoeducation, exposure, and cognitive-behavioral therapy, family-based treatment, or applied behavior analysis approaches. Occupational therapists assess and address feeding difficulties by considering sensory differences, physical and cognitive impairments, as well as broader contextual factors such as social environments, mealtime rituals and routines, culture, and social factors. It has been emphasized that occupational therapy interventions are needed for individuals with ARFID. Occupational therapists have demonstrated effectiveness using approaches such as the Sequential Oral Sensory (SOS) Feeding Approach, Sensory Integration, the Just Right Challenge Feeding Protocol, and family-based programs such as Occupational Performance Coaching (OPC). Studies highlight the need to standardize occupational therapy approaches for ARFID and to conduct single-case experimental designs and randomized controlled trials comparing these approaches with alternative methods.

In this context, the Sequential Oral Sensory (SOS) Feeding Approach is a structured intervention that supports sensory-motor skills related to feeding and aims to help the child develop a positive relationship with food. By gradually increasing interaction with food, the SOS approach aims to reduce sensory sensitivities and improve feeding behaviors. It has been shown to be effective particularly in children with autism spectrum disorder and in other diagnostic groups with feeding difficulties. However, no randomized controlled trial has yet been found addressing the use of this approach in children with ARFID.

On the other hand, Occupational Performance Coaching (OPC) is a structured, problem-solving, guidance, and empowerment-based approach designed to help parents support their children's daily life performance. Studies conducted with families of children with developmental differences have shown that OPC contributes positively to parental self-efficacy, stress levels, and children's participation levels. While studies have demonstrated its effectiveness in children with selective eating problems, it has been emphasized that its effectiveness should be further tested in randomized controlled trials.

Despite existing psychosocial interventions for ARFID, the literature highlights a lack of sensory- and behaviorally-oriented feeding interventions. Therefore, this randomized controlled single-blind study aims to examine the effects of the SOS approach alone and in combination with OPC on feeding problems and feeding behaviors of children with ARFID, as well as on parental feeding attitudes and mealtime behaviors. By going beyond child-focused sensory-based interventions, this study also evaluates the effectiveness of family-centered approaches. The study aims to make an original contribution to the development of applicable and effective intervention models for children and families dealing with ARFID, both at the clinical and societal levels.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria (for the child):

  * Having been diagnosed with ARFID according to the DSM-5 by a Child and Adolescent Mental Health and Diseases psychiatrist (Assoc. Prof. Dr. Hakan ÖĞÜTLÜ).
  * Being between the ages of 3 and 8.
  * Being medically stable for outpatient treatment.
  * Having no conditions (visual, auditory, cognitive, or chewing) that would prevent participation in treatment.

Inclusion Criteria (for the mother):

* Being the child's primary caregiver and living with the mother.
* Having at least a primary school diploma and possessing Turkish reading and comprehension proficiency.
* Agreeing to take an active role in the intervention process and participate in research evaluations.
* Being a regular participant in the child's feeding process.
* Not having another child with special needs.

Exclusion Criteria:

* Exclusion Criteria (Child):

  * History of comorbid neurological, genetic, psychiatric, or metabolic disease
  * Child and family receiving other individual or family-based education and/or psychotherapy during the intervention
  * Taking medication for comorbid disorders affecting appetite and/or weight
  * Active psychiatric crisis (e.g., severe anxiety disorder, post-traumatic stress disorder)
  * Significant family or environmental constraints that would prevent regular attendance

Exclusion Criteria (Mother):

* Severe hearing, vision, or cognitive impairment
* Child concurrent participation in another intervention program (dietician, psychotherapy, group education, etc.) related to feeding behaviors
* Presence of a chronic health condition (e.g., neurological, psychiatric, orthopedic, oncological, etc.) that would prevent regular attendance at the intervention

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Behavioral Pediatric Feeding Scale | 12 weeks
  The Behavioral Pediatric Feeding Assessment Scale (BPFAS), was adapted into Turkish , and later studied with parents of children aged 3-12 years attending preschool and primary school. The original scale consists of 35 items, 25 of which relate to the child's feeding behavior and 10 to the caregiver responsible for feeding. However, the Turkish adaptation was conducted using only the 25 items related to the child. Among these, six items are positively worded (items 1, 3, 5, 6, 9, and 16), while the remaining 19 are negatively worded. Responses are scored on a five-point Likert scale ranging from 1 (never) to 5 (always), with positively worded items reverse-scored. Parents are asked whether each item represents a problem for them. A total score above 84 indicates the presence of a feeding disorder, while reporting more than nine problematic items reflects a high number of feeding-r
Children's Eating Behavior Questionnaire | 12 weeks
  The Children's Eating Behaviour Questionnaire (CEBQ), is a parent-reported, Likert-type questionnaire designed to assess eating behaviors in children aged 2-9 years. It includes 35 items rated on a 5-point scale (1 = never, 5 = always) and encompasses eight subscales that reflect different aspects of children's eating behaviors. Reported Cronbach's alpha coefficients for the original scale range from 0.72 to 0.91, indicating good internal consistency. The validity and reliability of the CEBQ in Turkey were examined.The scale consists of eight subscales that can be grouped into two main dimensions.
Sensory Eating Problems Scale | 12 weeks
  The Sensory Eating Problems Scale (SEPS) was developed for children aged 3-11 years to evaluate sensory-related feeding difficulties. The scale consists of 22 items rated on a 5-point Likert scale (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = always) and includes six subscales: Food Texture Aversion, Single Food Focus, Vomiting, Temperature Sensitivity, Expulsion, and Overstuffing. SEPS is completed by the child's caregiver. Confirmatory factor analysis by Seiverling et al. (2019) reported χ²/df = 2.63, CFI = 0.90, and RMSEA = 0.06, supporting the six-factor model as an acceptable structure for assessing sensory feeding problems. In addition, Cronbach's alpha values for the subscales were 0.85 for Food Texture Aversion, 0.70 for Single Food Focus, 0.73 for Vomiting, 0.72 for Temperature Sensitivity, 0.71 for Expulsion, and 0.71 for Overstuffing. The Turkish validity and reliability study was conducted by Demirok et al. in children aged 3-11 years.
Sensory Profile | 12 weeks
  The Sensory Profile, developed by Dunn and colleagues, is used to assess sensory processing abilities in children aged 3-10 years. It consists of 125 items and evaluates three main domains: Sensory Processing (6 subdomains), Sensory Modulation (5 subdomains), and Behavioral and Emotional Responses (3 subdomains). The subdomains include Auditory Processing, Visual Processing, Vestibular Processing, Tactile Processing, Multisensory Processing, Oral Sensory Processing, Sensory Processing related to Endurance and Tone, Regulation of Movement and Body Position, Regulation of Activity Level by Movement, Modulation of Sensory Input Affecting Emotional Responses, Modulation of Visual Input Affecting Emotional Responses and Activity Level, Emotional/Social Responses, Behavioral Outcomes of Sensory Processing, and Items Indicating Thresholds of Responsiveness. The Turkish validity and reliability study of the scale was conducted by Kayıhan and colleagues.
Goal Attainment Scale (GAS) | 12 weeks
  The Goal Attainment Scaling (GAS) is widely used in patient-centered treatment approaches with no age restrictions, and it is based on the principle of collaboratively setting treatment goals between the therapist and the patient. In this study, parents are asked during the initial assessment to define five individual goals they wish to achieve throughout the therapy process. Each goal is prioritized by the parent, who also rates the perceived level of difficulty. At the post-treatment evaluation, each goal is scored on a five-point scale ranging from -2 to +2 (-2 = much less than expected outcome, -1 = somewhat less than expected, 0 = expected outcome, +1 = somewhat more than expected, +2 = much more than expected). As a performance-based measure, GAS does not require separate validity and reliability testing for the Turkish context.

SECONDARY OUTCOMES:
Parental Feeding Style Questionnaire | 12 weeks
  The Parent's Feeding Style Questionnaire (PFSQ), developed by Wardle et al. (2002), was adapted into Turkish by Özçetin et al. (2010) in a study including 468 parents of children aged 2-9 years. In the original version, the four-factor structure showed Cronbach's alpha values ranging from 0.67 to 0.85. In the Turkish validity and reliability study, a five-factor structure was identified, where the original "control over eating" factor was divided into "strict control feeding" and "permissive control feeding." Cronbach's alpha coefficients for the Turkish version ranged from 0.54 to 0.83 across the factors.
Maternal Attitudes towards the Feeding Process Scale | 12 weeks
  The mother's attitude during the feeding process was assessed using the Feeding Process Maternal Attitude Scale. The validity of this scale was tested in mothers over the age of 18. It consists of 27 items and five subscales. In this study, the internal consistency coefficient was found to be Cronbach's α = 0.88. The scale is rated on a five-point Likert system (1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always), with a minimum possible score of 27 and a maximum of 135. The subscales are: negative emotional state during meals, attitudes toward inadequate/unbalanced nutrition, negative feeding strategies, force-feeding, and reaction to others' opinions. Higher scores indicate an increase in problematic maternal attitudes related to the feeding process. Since the scale has no cut-off score, results were ranked from lowest to highest and divided into quartiles for evaluation.
Parenting Stress Index-Short Form | 12 weeks
  The Parenting Stress Index (PSI) was developed by Abidin (1982) to assess the level of stress experienced by parents of children with developmental disorders. The short form of the PSI (PSI-SF) was adapted into Turkish for parents of children aged 6 months to 14 years. The PSI-SF consists of 36 items across three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. In addition to subscale scores, a total stress score can also be calculated. Reported internal consistency (Cronbach's alpha) coefficients were 0.71 for the total stress score, 0.81 for the Parental Distress subscale (items 1-12), 0.76 for the Parent-Child Dysfunctional Interaction subscale (items 13-24), and 0.78 for the Difficult Child subscale (items 25-36). Test-retest reliability was reported as r = 0.88. Researchers have concluded that the scale is a suitable tool for measuring parenting stress and demonstrates cross-cultural validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Department of Occupational Therapy, Pediatric Unit, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data (IPD) that underlie the results reported in published articles, including de-identified demographic characteristics, baseline assessments, outcome measures, and intervention-related data. All shared IPD will be fully anonymized to ensure participant confidentiality.
Supporting Information: SAP, CSR
Time Frame: Individual participant data (IPD) and supporting documents will be available starting 6 months after publication of the primary study results and will remain accessible for 5 years thereafter.
Access Criteria: De-identified individual participant data (IPD) and supporting documents will be available to qualified researchers from academic institutions, hospitals, or recognized research organizations. Data will be shared only for projects with a sound scientific rationale and an established analysis plan. Researchers must submit a formal request describing study aims, methodology, and data protection procedures. Access will be granted through a secure, password-protected platform managed by the sponsor. Approved researchers will be required to sign a data use agreement to ensure confidentiality, proper use of the data, and compliance with ethical and legal standards.
URL: https://ergoterapi.hacettepe.edu.tr/tr/menu/akademik_personel-15

REFERENCES:
- [Background] Chilman LB, Meredith PJ, Southon N, Kennedy-Behr A, Frakking T, Swanepoel L, Verdonck M. Occupational Performance Coaching for parents of picky eaters: A mixed methods study. Aust Occup Ther J. 2024 Oct;71(5):644-660. doi: 10.1111/1440-1630.12947. Epub 2024 Mar 27. PMID 38538542
- [Background] Angelin CS, Sugi S, Rajendran K. Occupational Performance Coaching for Mothers of Children with Disabilities in India. Can J Occup Ther. 2021 Mar;88(1):38-47. doi: 10.1177/0008417420972868. Epub 2020 Dec 23. PMID 33353385
- [Background] Graham F. Occupational performance coaching: Client-centered and goal-directed practice; A commentary on collaborations with Sylvia Rodger. Aust Occup Ther J. 2017 Jul;64 Suppl 1:31-32. doi: 10.1111/1440-1630.12367. No abstract available. PMID 28714162
- [Result] Schoen SA, Balderrama R, Dopheide E, Harris A, Hoffman L, Sasse S. Methodological Components for Evaluating Intervention Effectiveness of SOS Feeding Approach: A Feasibility Study. Children (Basel). 2025 Mar 17;12(3):373. doi: 10.3390/children12030373. PMID 40150655
- [Result] Chilman LB, Meredith PJ, Kennedy-Behr A, Campbell G, Frakking T, Swanepoel L, Verdonck M. Picky eating in children: Current clinical trends, practices, and observations within the Australian health-care context. Aust Occup Ther J. 2023 Aug;70(4):471-486. doi: 10.1111/1440-1630.12869. Epub 2023 May 1. PMID 37127548
- [Result] Peterson KM, Piazza CC, Volkert VM. A comparison of a modified sequential oral sensory approach to an applied behavior-analytic approach in the treatment of food selectivity in children with autism spectrum disorder. J Appl Behav Anal. 2016 Sep;49(3):485-511. doi: 10.1002/jaba.332. Epub 2016 Jul 23. PMID 27449267
- See also: About OPC — https://www.scribd.com/document/619272118/Occupational-Performance-Coaching
- See also: About SOS — https://sosapproachtofeeding.com/